CLINICAL TRIAL: NCT01788241
Title: A Psycho-biochemical Perspective on Non-significant Coronary Artery Disease: a Prospective Cohort Study of Classic and Novel Risk Markers.
Brief Title: TweeSteden Mild Stenosis Study
Acronym: TWIST
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tilburg University (Other)
Collaborators: The Elisabeth-TweeSteden Hospital (Other); Elisabeth-TweeSteden Ziekenhuis (Other)
Responsible Party: Principal Investigator, Paula M.C. Mommersteeg, Assistant Professor, Tilburg University
Other Study IDs: UVT-MP-003
Record Dates: First submitted 2013-01-30; First posted 2013-02-11 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Coronary Artery Disease; Non-significant Coronary Artery Disease; Mild Stenosis; Vascular Irregularities
Keywords: coronary artery disease; Atherosclerosis; Coronary Stenosis; Cardiovascular Diseases; Non-significant coronary artery disease; Mild Stenosis; Vascular Irregularities; Psychosocial factors; Personality; Type D personality; Hostility; Depression; Anxiety; Fatigue; Social Support; Socioeconomic Status; Patient Reported Outcomes; Patient Perceived Symptoms; Health Status; Quality of Life; Chest pain; Cardiac risk factors; Metabolic Syndrome; BMI; Obesity; Waist Circumference; Lifestyle; Smoking; Alcohol use; Activity; Hypertension; Diabetes; Familial Cardiovascular Disease; Coronary angiography; Computed Tomography
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Coronary Stenosis; Cardiovascular Diseases; Depression; Anxiety Disorders; Fatigue; Chest Pain; Metabolic Syndrome; Obesity; Smoking; Alcohol Drinking; Motor Activity; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, DNA, leukocyte differentiation, high-sensitive C-reactive protein, fibrinogen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CAG and CT group: CAG group = patients included based on coronary angiography screening; CT group = patients included based on computed tomography screening

SUMMARY:
Psychosocial factors have been found to be associated with an increased risk for coronary artery disease incidence, progression and worse clinical outcomes.

Patients with non-significant coronary artery disease (confirmed vascular irregularities, but <60% coronary occlusion) often present with complaints such as chest pain, which warrant screening by coronary angiography (CAG) or computed tomography (CT scan). The prognosis of this group of patients with mild stenosis remains to be investigated in more detail, and we propose that psychosocial factors play a role in the clinical prognosis and patient reported outcomes in this group.

A special focus lies within examining personality characteristics, of which Type D personality is a primary predictor variable for prognosis. Type D personality is characterised by high negative affect and high social inhibition. In addition to psychosocial factors (personality, mood state, social support, SES), biomarkers(inflammation, clotting, DNA) as well as standard clinical risk factors (metabolic syndrome, activity level, smoking, medication use, disease severity) will be investigated.

The goal of the proposed study is to investigate a preexisting psycho-biochemical risk profile for major adverse cardiovascular events (MACE) and patient perceived symptoms in a group with angiographically or CT-scan confirmed, non-significant coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Based on quantitative coronary angiography (CAG): visible, but non-significant (<60% coronary occlusion) vascular irregularities and mild coronary stenosis.
* Based on 64-slice CT-scan (CT-scan): detected non-significant stenosis (calcium score >= lowest 10th percentile), and not eligible for CAG.

Exclusion Criteria:

* Normal coronary arteries (based on CAG or CT scan)
* Significant occlusion of coronary arteries (>=60% stenosis)
* Eligible for coronary intervention such as PCI or CABG
* History of coronary events (being either MI,PCI, CABG, heart failure)
* For the CT-screened group: eligible for CAG based on the CT-scan
* Serious comorbid conditions such as chronic kidney failure, or receiving chemotherapy
* Insufficient knowledge of the Dutch language

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have received coronary angiography or computed tomography at the TweeSteden Hospital Tilburg are being screened since January 2009.
Sampling Method: Probability Sample
Enrollment: 547 (Actual)
Dates: Start 2009-01; Primary Completion 2015-04 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | Average 42 months (Range 12-72; at least 12 months after inclusion final participant)
  MACE includes the occurence of a recurrent coronary angiography, emergency hospitalization (for cardiac reasons), myocardial infarction, percutaneous coronary intervention (PCI) or coronary artery bypass graft surgery (CABG), mortality (cardiac/noncardiac)
Patient Perceived Health Status | 12 and 24 months
  patient perceived health status includes self-reported chest pain, disease specific health status, generic health status, fatigue and mood (depression/anxiety). Double time point was included for this outcome measure to examine changes over time, compared to baseline.

SECONDARY OUTCOMES:
Psychosocial factors | baseline, 12 and 24 months
  The secondary aim is to investigate the correlation and the stability over time between psychosocial factors, biochemical variables, traditional cardiac risk factors and measures of outcome.
  Psychosocial factors include questionnaires as personality scales (Type D personality, Cook-Medley Hostility scale 27 item version), depression (HADS-D at each time point, BDI, CESD-10 and PHQ9 at consecutive time points), anxiety (HADS-A at each time point), fatigue (FAS), global mood scale (Positive and negative affect), generic health status (Short Form 12), specific health status (Seattle Angina Questionnaire). Indicators of education level, marital status, lifestyle factors, and activity level.
Biochemical correlates | baseline, 12 and 24 months
  Examine biochemical correlates in relation to psychosocial and traditional cardiac risk factors.
  Standard assessment is done for high sensitive C-reactive protein (hsCRP), fibrinogen, leukocyte count and differentiation, and registration of lipid profile, glucose, creatinin at baseline. Baseline and 12 month serum samples are collected and stored at -80, as well as DNA samples for future funding opportunities.

CONTACTS AND LOCATIONS:
Overall Officials: Paula M.C. Mommersteeg, PhD, Principal Investigator — Tilburg University; Jos W. Widdershoven, MD PhD, Principal Investigator — The Elisabeth-TweeSteden Hospital; Wilbert Aarnoudse, MD PhD, Study Chair — The Elisabeth-TweeSteden Hospital; Johan Denollet, PhD, Study Chair — Tilburg University
Locations (1):
- TweeSteden Hospital Tilburg, Tilburg, Dr. Deelenlaan 5, Netherlands

REFERENCES:
- [Result] Mommersteeg PM, Pot I, Aarnoudse W, Denollet J, Widdershoven JW. Type D personality and patient-perceived health in nonsignificant coronary artery disease: the TWeesteden mIld STenosis (TWIST) study. Qual Life Res. 2013 Oct;22(8):2041-50. doi: 10.1007/s11136-012-0340-2. Epub 2012 Dec 21. PMID 23263915
- [Result] Mommersteeg PM, Meeuwis SH, Denollet J, Widdershoven JW, Aarnoudse W, Westerhuis BL, Kop WJ. C-reactive protein and fibrinogen in non-obstructive coronary artery disease as related to depressive symptoms and anxiety: findings from the TweeSteden Mild Stenosis Study (TWIST). J Psychosom Res. 2014 Nov;77(5):426-9. doi: 10.1016/j.jpsychores.2014.09.020. Epub 2014 Oct 2. PMID 25307791
- [Result] Mommersteeg PM, Widdershoven JW, Aarnoudse W, Denollet J. Personality subtypes and chest pain in patients with nonobstructive coronary artery disease from the TweeSteden Mild Stenosis study: mediating effect of anxiety and depression. Eur J Pain. 2016 Mar;20(3):427-37. doi: 10.1002/ejp.743. Epub 2015 Jun 24. PMID 26105088
- [Derived] Mommersteeg PMC, Naude PJW, Bagijn W, Widdershoven J, Westerhuis BWJJM, Schoemaker RG. Gender differences in associations of depressive symptoms and anxiety with inflammatory markers in patients with non-obstructive coronary artery disease. J Psychosom Res. 2019 Oct;125:109779. doi: 10.1016/j.jpsychores.2019.109779. Epub 2019 Jul 17. PMID 31421324
- [Derived] Mommersteeg PM, Arts L, Zijlstra W, Widdershoven JW, Aarnoudse W, Denollet J. Impaired Health Status, Psychological Distress, and Personality in Women and Men With Nonobstructive Coronary Artery Disease: Sex and Gender Differences: The TWIST (Tweesteden Mild Stenosis) Study. Circ Cardiovasc Qual Outcomes. 2017 Feb;10(2):e003387. doi: 10.1161/CIRCOUTCOMES.116.003387. Epub 2017 Feb 22. PMID 28228453
- See also: CoRPS: Center of Research on Psychology in Somatic diseases. Primary funding for the TWIST study. — http://www.tilburguniversity.edu/research/institutes-and-research-groups/corps/
- See also: TweeSteden Hospital, Tilburg, the Netherlands. Study location and CoRPS collaboration [Site in Dutch] — https://www.tweestedenziekenhuis.nl/